CLINICAL TRIAL: NCT03254914
Title: A Multi-center, Cluster-randomized, Prospective, Observational Study
Brief Title: Fimasartan Optimal Reduction Targeting Elevated Blood Pressure: the FORTE Study
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-FMS-OS-403
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hypertension
Keywords: Home Blood Pressure; Fimasartan
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Site: Measure Clinic Blood Pressure
- Test Site: Measure Clinic Blood Pressure and Home Blood Pressure
  Interventions: Procedure: Home Blood Pressure

INTERVENTIONS:
Procedure: Home Blood Pressure — Measure Home Blood Pressure
  Groups: Test Site

SUMMARY:
The purpose of this study is to evaluate the effect of home blood pressure monitoring on controlling blood pressure and correlation between home blood pressure and clinic blood pressure in hypertensive patients receiving two or more concomitant antihypertensive agents including fimasartan

DETAILED DESCRIPTION:
A multi-center, cluster-randomized, prospective, observational study

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily signed informed consent for participating in this clinical study
* Male and female over the age of 19
* Hypertensive patients receiving two or more concomitant anti-hypertensive agents including fimasartan

Exclusion Criteria:

* Renal dialysis patients.
* Diabetic nephropathy patients taking angiotensin-converting enzyme inhibitor.
* Severe renal disorder
* Subjects with hereditary disorders of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* Medical history with hypersensitivity to Fimasartan
* Pregnant women or lactating female.
* Participate in another clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients
Sampling Method: Non-Probability Sample
Enrollment: 3554 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Rate of reaching target blood pressure | 12 weeks after treatment
  Rate of reaching target blood pressure after treatment for 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi JY, Kim KI, Kim CH. Effect of home blood pressure monitoring for blood pressure control in hypertensive patients taking multiple antihypertensive medications including fimasartan (the FORTE study). Clin Hypertens. 2020 Dec 15;26(1):24. doi: 10.1186/s40885-020-00154-y. PMID 33317628